CLINICAL TRIAL: NCT01064037
Title: A Placebo Controlled, Randomized, Double-Blind, Fixed-dose, Multicenter, Phase IIb Study to Investigate the Efficacy and Tolerability of BAY 58-2667 (50 µg/h, 100 µg/h, 150 µg/h) Given Intravenously to Subjects With Acute Decompensated Chronic Congestive Heart Failure (ADHF) Within 12 Hours After Hospital Admission (Pulmonary Artery Catheter eg, Swan-Ganz Not Required)
Brief Title: A Phase IIb Study to Investigate the Efficacy and Tolerability of Cinaciguat (150 µg/h, 100 µg/h, 50 µg/h) Given Intravenously to Subjects With Acute Decompensated Chronic Congestive Heart Failure (ADHF)
Acronym: COMPOSE EARLY
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14836; 2009-017082-39 (EudraCT Number)
Record Dates: First submitted 2010-02-04; First posted 2010-02-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Heart Failure; Heart Decompensation
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — BAY 58-2667

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: Cinaciguat (BAY58-2667)
- Arm 2 (Experimental)
  Interventions: Drug: Cinaciguat (BAY58-2667)
- Arm 3 (Experimental)
  Interventions: Drug: Cinaciguat (BAY58-2667)
- Arm 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cinaciguat (BAY58-2667) — Infusion of 150 µg/h during 48h.
  Arms: Arm 1
Drug: Cinaciguat (BAY58-2667) — Infusion of 100 µg/h during 48h
  Arms: Arm 2
Drug: Cinaciguat (BAY58-2667) — Infusion of 50 µg/h during 48h
  Arms: Arm 3
Drug: Placebo — Infusion during 48h
  Arms: Arm 4

SUMMARY:
A placebo controlled, double-blind and randomized study to assess different doses of a new drug (BAY58-2667) given intravenously, to evaluate if it is safe and can help to improve the well-being of patients with acute decompensated heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant, non-lactating female subjects, age >/= 18 years of age; or women without childbearing potential defined as postmenopausal women aged 55 years or older, women with bilateral tubal ligation, women with bilateral ovarectomy, and women with a hysterectomy
* Subjects must have the clinical diagnosis of congestive heart failure (CHF) made at least three months prior to enrollment
* Subjects must experience worsening of both of the symptoms below leading to hospitalization at the time of entry into the study: dyspnea and clinical evidence of volume overload

Exclusion Criteria:

* Acute de-novo heart failure
* Acute myocardial infarction and/or myocardial infarction within 30 days
* Valvular heart disease requiring surgical intervention during the course of the study
* Heart failure due to or associated with uncorrected primary valvular disease, malfunctioning artificial heart valve, or uncorrected congenital heart disease
* Primary hypertrophic cardiomyopathy
* Acute inflammatory heart disease, eg, acute myocarditis
* Unstable angina requiring angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-04; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Dyspnea VAS (using a visual analogue scale) | 8 hours

SECONDARY OUTCOMES:
Dyspnea assessment (Likert Scale) | up to follow-up (30 - 35 days)
Overall health status assessment (EQ-5D) | up to follow-up (30 - 35 days)
Changes in the dyspnea VAS at other time points | Up to follow up visit
Dyspnea assessment through Likert scale | Up to follow up visit
Overall health status assessment through EQ-5D Health Questionnaire | Up to the follow-up visit
Global clinical assessment by the physician | At 8, 24, and 48 hours
Change in concomitant medications | During the treatment
Safety variables | Up to end of study
  Frequency of TEAEs (AEs were considered to be treatment emergent if they started after the start of sthe study drug infusion to up to 2 calendar days after the end of the study drug infusion); treatment-emergent serious adverse events (SAEs); deaths; evaluation of renal and cardiac function; Change in heart rate; Change in systolic and diastolic blood pressure; Laboratory parameters (including parameters related to hematology, clinical chemistry, urinalysis, and biomarkers); ECG assessment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (62):
- United States (6):
  - Chicago, Illinois
  - Detroit, Michigan
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Nashville, Tennessee
  - Houston, Texas
- Canada (3):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Québec, Quebec
- Czechia (3):
  - Brno
  - Pardubice
  - Prague
- Finland (2):
  - Jyväskylä, Jyväskylä
  - Turku, Turku
- France (3):
  - Dommartin-lès-Toul
  - Paris
  - Poitiers
- Germany (6):
  - Nuremberg, Bavaria
  - Melsungen, Hesse
  - Mönchengladbach, North Rhine-Westphalia
  - Kiel, Schleswig-Holstein
  - Berlin, State of Berlin
  - Erfurt, Thuringia
- Hungary (3):
  - Budapest
  - Kecskemét
  - Székesfehérvár
- Ireland (3):
  - Ballinasloe, Co. Galway
  - Dublin, Dublin
  - Dublin
- Israel (4):
  - Haifa, Israel
  - Rehovot, Israel
  - Safed, Israel
  - Nahariya
- Italy (7):
  - Pontedecimo, Genova
  - Casarano, Lecce
  - Cotignola, Ravenna
  - Bari
  - Ferrara
  - Padua
  - Roma
- Japan (7):
  - Kanazawa, Ishikawa-ken
  - Kagoshima, Kagoshima-ken
  - Chigasaki, Kanagawa
  - Matsumoto, Nagano
  - Shizuoka, Shizuoka
  - Sunto, Shizuoka
  - Tanabe, Wakayama
- Poland (4):
  - Bydgoszcz
  - Krakow
  - Olsztyn
  - Szczecin
- South Africa (3):
  - Johannesburg, Gauteng
  - Kuils River, Western Cape
  - Worcester, Western Cape
- South Korea (2):
  - Seoul, Jongno-gu,
  - Seoul, Songpa-gu
- Spain (4):
  - Torrevieja, Alicante
  - Barcelona, Barcelona
  - Majadahonda, Madrid
  - El Palmar, Murcia
- United Kingdom (2):
  - Harrow, London
  - Northampton, Northamptonshire

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/